CLINICAL TRIAL: NCT05486234
Title: Brief Computerized Intervention for Reducing Adolescent Cannabis and Alcohol Use
Brief Title: CARS: Cannabis and Alcohol Reduction Study
Acronym: CARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00106723; 1K23DA050800-01A1 (NIH)
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use; Alcohol Use, Unspecified; Substance Use; Substance Use Disorders
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Treatment Group (Experimental)
  Interventions: Behavioral: modified Approach-Avoidance Task (mAAT), which aims to modify automatic approach bias
- Group B: Control Group (Sham Comparator)
  Interventions: Behavioral: modified Approach-Avoidance Task (mAAT) that does not aim to modify automatic approach bias.

INTERVENTIONS:
Behavioral: modified Approach-Avoidance Task (mAAT), which aims to modify automatic approach bias — Participants will undergo a baseline assessment before completing computerized tasks. During the baseline assessment, participants will be asked questions about alcohol and cannabis use. We will also ask questions about the way participants think about things, past life experiences related to substance use, and questions about how participants feel about reducing their substance use. Then, participants will complete a series computerized tasks where they will push and pull a joystick in response to images that are presented on a screen or where they will try to get a high score. During the computerized tasks, we will also be measuring brain activity using EEG. During the study, participants will also be asked to respond to questions about their health and behavior using an app on a smartphone or tablet using a secure program. Participants in the Treatment Group will then complete four sessions of the modified Approach-Avoidance Task (mAAT), which aims to modify automatic approach bias.
  Arms: Group A: Treatment Group
Behavioral: modified Approach-Avoidance Task (mAAT) that does not aim to modify automatic approach bias. — Participants will undergo a baseline assessment before completing computerized tasks. During the baseline assessment, participants will be asked questions about alcohol and cannabis use. We will also ask questions about the way participants think about things, past life experiences related to substance use, and questions about how participants feel about reducing their substance use. Then, participants will complete a series computerized tasks where they will push and pull a joystick in response to images that are presented on a screen or where they will try to get a high score. During the computerized tasks, we will also be measuring brain activity using EEG. During the study, participants will also be asked to respond to questions about their health and behavior using an app on a smartphone or tablet using a secure program. Participants in the Control Group will then complete four sessions of an Approach-Avoidance Task (mAAT) that does not aim to modify automatic approach bias.
  Arms: Group B: Control Group

SUMMARY:
The study will test a computerized treatment with subjects ages 13-17 years who are seeking treatment for alcohol and/or cannabis use. Follow-up assessments will be conducted at one- and three-months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 13 and 17
* be seeking treatment for either cannabis or alcohol use;
* report co-occurring alcohol and cannabis use during the past three months (i.e., participants who report using both alcohol and cannabis during the three months prior to participation in the study, regardless of if the use was simultaneous)
* have a caregiver willing to participate and provide consent.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis use as assessed by Timeline Followback | Baseline and Three-Month Follow-up
  The TLFB is a calendar-assisted semi-structured interview that will be used to assess cannabis and alcohol use since the last assessment. The TLFB will assess the number of days a person used cannabis over the past 90 days compared to the 90 days prior to enrolling in this study.
Change in alcohol use as assessed by Timeline Followback | Baseline and Three-Month Follow-up
  The TLFB is a calendar-assisted semi-structured interview that will be used to assess cannabis and alcohol use since the last assessment. The TLFB will assess the number of days a person consumed alcohol over the past 90 days compared to the 90 days prior to enrolling in this study.
Change in Cannabis Approach Bias (D-Score) | Baseline, One-Week Follow-up, and Three-Month Follow-up
  D scores will be calculated for each participant at baseline, posttest, and three-month follow-up. Participants' mean reaction times (RTs) during the approach cannabis trials will be subtracted from the mean avoid cannabis trial RTs. These scores are then divided by the SD across all cannabis trials. Positive scores indicate an approach bias for cannabis stimuli.
Change Cannabis Approach Bias (D-Score) | Baseline, One-Week Follow-up, and Three-Month Follow-up
  D scores will be calculated for each participant at baseline, posttest, and three-month follow-up. Participants' mean reaction times (RTs) during the approach alcohol trials will be subtracted from the mean avoid alcohol trial RTs. These scores are then divided by the SD across all alcohol trials. Positive scores indicate an approach bias for alcohol stimuli.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No